CLINICAL TRIAL: NCT01614418
Title: Endoscopic Radiofrequency Ablation for Gastric Metaplasia and Dysplasia
Brief Title: Radiofrequency Ablation for Gastric Metaplasia and Dysplasia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, LEUNG Wai Keung, Clinical Professor, The University of Hong Kong
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HKU_WKL_RFA1
Record Dates: First submitted 2012-06-04; First posted 2012-06-08 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Gastric Dysplasia; Intestinal Metaplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endoscopic radiofrequency ablation (Experimental): Endoscopic radiofrequency ablation using BARRX HALO90 catheter
  Interventions: Device: Endoscopic radiofrequency ablation catheter

INTERVENTIONS:
Device: Endoscopic radiofrequency ablation catheter — Endoscopic radiofrequency ablation
  Other Names: BARRX HALO90

SUMMARY:
Gastric intestinal metaplasia (IM) and dysplasia, also referred to as intra-epithelial neoplasia, are well recognized precursors of gastric cancer. Apart from endoscopic surveillance, there is no other intervention which predictably eradicates pre-cancerous gastric lesions.

Endoscopic radiofrequency ablative (RFA) therapy has been recently shown to be highly effective in eradicating both IM and dysplasia in patients with Barrett's esophagus. However, the potential role of RFA to remove gastric IM and dysplasia remains unknown. In this study, we determine the feasibility of using endoscopic RFA in treating early gastric neoplasia (metaplasia and dysplasia). Patients with gastric metaplasia and/or dysplasia will be treated with endoscopic RFA. The safety and effects of RFA will be determined.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmation of gastric IM or dysplasia.
2. The lesion is no larger than 5 cm in diameter.
3. Age ≥ 18 years.
4. No previous endoscopic mucosal resection or submucosal dissection.
5. No active H. pylori infection.
6. Subject is able to tolerate endoscopy and sedation.
7. Subject agrees to participate, fully understands content of the informed consent, and signs the informed consent form.

Exclusion Criteria:

1. Gastric cancer (intra-mucosal cancer or worse).
2. Prior gastric irradiation or surgery.
3. Anti-platelet or anti-thrombotic medication use that cannot be stopped for 7 days before and after RFA.
4. Gastric ulcers, fistulae and varices.
5. History of alcohol and/or controlled substance dependency.
6. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Histological clearance of dysplasia/metaplasia | 6 month

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | up to 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Wai Keung Leung, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Leung WK, Tong DK, Leung SY, Chan FS, Tong TS, Ho RS, Chu KM, Law SY. Treatment of Gastric Metaplasia or Dysplasia by Endoscopic Radiofrequency Ablation: A Pilot Study. Hepatogastroenterology. 2015 May;62(139):748-51. PMID 26897966